CLINICAL TRIAL: NCT06050434
Title: PROTraSarc Prospective Study to Evaluate Patient Reported Outcomes (PRO) During Rechallenge With Trabectedin in Sarcoma Patients - A GISAR Sub-study
Brief Title: Prospective Study to Evaluate Patient Reported Outcomes (PRO) During Rechallenge With Trabectedin in Sarcoma Patients
Acronym: PROTraSarc
Status: Terminated | Type: Observational
Why Stopped: The study was terminated prematurely due to slow recruitment after inclusion of 7 patients (of initially planned 100 patients).
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Collaborators: PharmaMar (Industry)
Responsible Party: Sponsor
Other Study IDs: PROTraSarc
Record Dates: First submitted 2023-07-12; First posted 2023-09-22 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Soft Tissue Sarcoma
Keywords: Re-Challenge; Trabectedin; Sarcoma; registry; PRO
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trabectedin Rechallenge in Soft sarcoma patients: Adult GISAR participants with Trabectedin-pretreated soft tissue sarcomas and rechallenge with at least one cycle of Trabectedin in any line of therapy, with the interval between Trabectedin interruption and Trabectedin rechallenge being at least 3 months.

SUMMARY:
Chemotherapy with Trabectedin is an effective treatment for sarcoma patients in the second line setting or in first line for patients who are deemed unsuitable to receive anthracycline therapy. The prospective study will primarily investigate the PRO of Trabectedin rechallenge in patients with soft tissue sarcomas that had to discontinue initial Trabectedin treatment due to various reasons such as progression, side effects or surgery, as is commonly the case in real-life settings. Embedding this trial in the GISAR registry enables the evaluation of a large number of patients with long-term follow-up which allows multiple analyses regarding different questions that remain unanswered until today.

DETAILED DESCRIPTION:
Chemotherapy with Trabectedin is an effective treatment for sarcoma patients in the second line setting or in first line for patients who are deemed unsuitable to receive anthracycline therapy. Several features differentiate its clinical performance from other chemotherapeutic agents, including durability of response and the absence of cumulative toxicity even upon re-exposition to treatment after interruption of therapy. In addition, the results of the T-Dis trial evaluating the impact of Trabectedin rechallenge demonstrated that it retains its activity when patients are rechallenged on progression after a treatment break.

Since sarcoma patient usually report a worse global quality of life (QoL) compared to the general population, one of the main goals of treating advanced-stage patients with Trabectedin, in addition to its efficacy, is to improve the QoL, represented by symptom control and other patient-related outcomes. However, little is known to date about the QoL during a rechallenge with Trabectedin, after patients had to discontinue Trabectedin treatment.

Patient-reported outcome (PRO) measures are standardized questionnaires that collect information on health outcomes directly from the patients, including symptoms, health-related QoL parameters and functional status. In general, there are two types of PROMs, disease-specific and general measures that can also be used for healthy populations. A growing number of articles supports the need for, as well as the benefit of, deriving information directly from patients. Thus, the application of PRO measures, initially developed for the use in research, has become more common nowadays and their application is included in supporting clinical decision making, comparing outcomes among health-care providers, stimulating quality improvement and evaluating practices and policies. Therefore, the collection of real-world data from patients subject to Trabectedin rechallenge would enable further estimations on the feasibility and efficacy of Trabectedin rechallenge.

The prospective PROTraSarc sub-study will primarily investigate the PRO of Trabectedin rechallenge in patients with soft tissue sarcomas that had to discontinue initial Trabectedin treatment due to various reasons such as progression, side effects or surgery, as is commonly the case in real-life settings. Embedding this trial in the GISAR registry enables the evaluation of a large number of patients with long-term follow-up which allows multiple analyses regarding different questions that remain unanswered until today.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled participant of the GISAR registry and their sub-studies
* Patient with histologically confirmed soft tissue sarcomas
* Pretreatment with Trabectedin, termination of this therapy regardless of reason
* Planned rechallenge or started rechallenge with Trabectedin in any line of therapy within 2 weeks before inclusion
* Interval between last Trabectedin treatment and Trabectedin rechallenge at least 3 months

Exclusion Criteria:

* Not able to understand all implications of study participation
* No written informed consent
* Age ≤ 18 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult GISAR participants with Trabectedin-pretreated soft tissue sarcomas and rechallenge with at least one cycle of Trabectedin in any line of therapy, with the interval between Trabectedin interruption and Trabectedin rechallenge being at least 3 months.
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2023-10-31 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Patient reported outcome regarding symptoms and side effects during Trabectedin re-challenge in soft tissue sarcoma patients | through study completion, an average of 2 years
  PRO-CTCAE questionnaire
Patient reported outcome regarding distress during Trabectedin re-challenge in soft tissue sarcoma patients | through study completion, an average of 2 years
  Distress-Thermometer
Patient reported outcome regarding quality of life during Trabectedin re-challenge in soft tissue sarcoma patients | through study completion, an average of 2 years
  QLQ-C30 Questionnaire
Patient reported outcome regarding cancer behaviour inventory | every nine to 18 weeks during Trabectedin re-challenge, every 3 Month in follow up
  CBI-B Questionnaire
Patient reported outcome measuring anxiety and depression | through study completion, an average of 2 years
  PHQ-4 Questionnaire
Patient reported outcome measuring self-efficacy for managing chronic disease | through study completion, an average of 2 years
  SES6G Questionnaire

SECONDARY OUTCOMES:
Analysis of correlation of PROs with clinical parameters | through study completion, an average of 2 years
  Evaluation of different PROs and analysis of correlation with clinical parameters, e.g. therapy response and side effects experienced during therapy
Characterization of patients receiving Trabectedin rechallenge in real life setting | through study completion, an average of 2 years
  Characterization of patients receiving Trabectedin rechallenge in real life setting, e.g. demographics, previous therapies
Characterization of Trabectedin rechallenge in real life conditions | through study completion, an average of 2 years
  Characterization of Trabectedin rechallenge in real life conditions, e.g. number of Trabectedin cycles applied, response to therapy, reason for end of Trabectedin rechallenge (e.g. disease progression, intolerable toxicity, death)

OTHER OUTCOMES:
Assessment of PRO data capture via an electronic tool (ePRO) | through study completion, an average of 2 years
  Assessment of PRO data capture via an electronic tool (ePRO), e.g. handling, user experience, completion rate, adherence) and its implementation into the routine sarcoma patient care (parameters will e.g. include patient acceptance, represented by the rate of patients entering an ePRO tool at least once) for sarcoma patients under Trabectedin rechallenge

CONTACTS AND LOCATIONS:
Overall Officials: Markus Schuler, PD Dr. med., Principal Investigator — Onkologischer Schwerpunkt Oskar-Helene-Heim, Clinic and Polyclinic for Internal Medicine I, University Hospital Carl Gustav Carus, TU Dresden, Dresden, Germany; Daniel Pink, PD Dr. med., Principal Investigator — Sarcoma Center Berlin-Brandenburg, Helios Hospital Bad Saarow, Department of Internal Medicine C, University Hospital Greifswald, Germany; Salah-Eddin Al-Batran, Prof. Dr. med., Study Director — Institut für Klinische Krebsforschung am Krankenhaus Nordwest
Locations (9):
- Germany (9):
  - HELIOS KLinikum Bad Saarow, Bad Saarow
  - HELIOS Klinikum Berlin Buch, Berlin
  - Frankfurt Universitätsklinikum, Frankfurt am Main
  - Universitätsmedizin Göttingen, Göttingen
  - Universitätsmedizin Greifswald, Greifswald
  - Uniklinikum Leipzig, Leipzig
  - Universitätsmedizin Mainz, Mainz
  - Westfälische Wilhelms-Universität Münster, Münster
  - Universitätsklinikum Tübingen, Tübingen

IPD SHARING:
Plan to Share IPD: No
will not be shared